CLINICAL TRIAL: NCT04540198
Title: GamePlan4Care: Web-based Delivery System for REACH II
Brief Title: GamePlan4Care: Online Support for Family Caregivers
Acronym: GP4C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 018-622; R01AG061973-01 (NIH)
Record Dates: First submitted 2019-01-02; First posted 2020-09-07 (Actual); Results first posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2022-10

CONDITIONS: Dementia
Keywords: Caregiving; Skills-training
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GamePlan4Care (GP4C) (Experimental): Participants in this arm will have access to full functionality and content of the online system GamePlan4Care (GP4C) including educational resources, skills training, and support tailored to their unique caregiving needs. Additional individualized feedback will be automatically generated based on responses to online questions and will include links to relevant site educational/skill-building content. Participants will be assigned a Dementia Care Specialist who will facilitate caregiver interactions with the online material and provide skills training via telephone or web-video conference. Study participants assigned to GP4C will receive 9 automated emails and 4 phone calls over a 6-month period.
  Interventions: Behavioral: GamePlan4Care
- Resources4Care (R4C) (Active Comparator): Participants in this arm will receive access to Resources4Care (R4C), a feature-limited version GamePlan4Care system. R4C will serve as an online hub for articles and videos about Alzheimer's disease and dementia. Educational topics will included information on: 1) Alzheimer's Disease & Dementia, 2) Caregiving, 3) Caregiver Stress and 4) Home Safety. R4C will present a page on each topic with active links to two additional online sources on the same topic. Study participants assigned to R4C will receive two emails from their DCS encouraging the caregiver to review specific education materials. Each email will be followed by brief "check-in" calls (15-min each) at three months and five months after randomization.
  Interventions: Behavioral: Resources4Care

INTERVENTIONS:
Behavioral: GamePlan4Care — GamePlan4Care; Experimental
  Arms: GamePlan4Care (GP4C)
Behavioral: Resources4Care — R4C; Active Comparator
  Arms: Resources4Care (R4C)

SUMMARY:
As the population of older adults grows, almost doubling in size from 2012 to 2040, so too will the need for family caregiving. Caregiving can lead to negative psychosocial outcomes such as depression, anxiety, and burden; social isolation and family conflict: financial strain due to costs of care; and some caregivers also experience negative health consequences. This project will test the value of GamePlan4Care (GP4C) an evidence-based, internet-enabled system capable of providing immediate, tailored education and skills training to caregivers who can access live support from a DCS via phone or web-based video.

DETAILED DESCRIPTION:
Daily care and supervision of a person living with dementia (PWD) has been defined as "intense caregiving" and is associated with significant daily burdens and an overall threat to the caregiver's quality of life. Despite evidence suggesting that negative consequence can be remediated with community-based supports, those services remain allusive to caregivers due to the systemic challenges of turning interventions into services. This study is based on a practical approach of applying technology to an existing evidence-based intervention, Resources for Enhancing Alzheimer's Caregiver Health II (REACH II), refined with real-world user feedback and rigorously tested with the goal of creating an online family caregiver support system that has the potential of both scalability and sustainability. This two-group randomized controlled trial will compare the relative impact of GP4C to an education-based online site called Resources4Care (R4C) on a wide range of family caregiver outcomes. Family caregivers will be randomized to one of the two conditions and will complete an assessment battery at baseline and at the 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Must be age 18 years or older
* Providing at least 8 hours of weekly care and/or supervision (on average) for a friend or family member with a self-reported diagnosis of Alzheimer's disease or a related dementia. Family will be subjectively determined by the caregiver to enable a broader definition of a" "family" member often found in minority communities (e.g., a person not related by blood but who serves in the role of an "aunt" or "grandchild").
* The family member, named as the care recipient (CR) in this proposal, must be diagnosed with AD/ADRD (self-report from the caregiver accepted) and is experiencing signs of dementia as verified by the family caregiver on the AD8 informant interview. A score of 2 or greater is the inclusion criteria.
* Must demonstrate access to a home computer with internet access to research staff and report using the computer to access the internet at least three times per week, on average.
* English-speaking caregivers
* Must reside within the recruitment area (Target counties within Texas: Bastrop, Bell, Blanco, Burnet, Caldwell, Coryell, Fayette, Hamilton, Hays, Lampasas, Lee, Llano, Milam, Mills, San Saba, Travis, Williamson)

Exclusion Criteria:

* Current participation in another caregiving evidence-based program
* Previous participation in usability testing for current system development

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2024-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan B Stevens, PhD, Principal Investigator — Baylor Research Institute
Locations (1):
- Alzheimer's Texas, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD for all the primary and secondary outcomes will be shared with outside investigators, after review and approval for data use requests. Data for potential collaborators will be compiled as de-identified datasets to safeguard participant confidentiality. We will make a standardized dataset available to approved investigators, based on a subset of data from the study database; this dataset will be compiled and available after completion of the the study.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available after a reasonable time has elapsed to allow the original investigators time to publish results. Upon completion of all planned analyses, data will be archived according to NIH policy.

REFERENCES:
- [Derived] Stevens AB, Cho J, Birchfield T, Reese J, Han G, Thorud JL, Ory MG. A randomized trial of two online platforms for dementia family caregivers: GamePlan4Care and Resources4Care. Alzheimers Dement. 2025 Oct;21(10):e70690. doi: 10.1002/alz.70690. PMID 41085219

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from various locations in Central Texas, including community-based organizations like Area Agencies on Aging and Alzheimer's nonprofits. Health system providers also referred family caregivers of patients diagnosed with dementia. This multi-faceted approach aimed to reach a diverse population of caregivers, enhancing the study's representativeness and engagement.
Pre-assignment Details: After participants expressed interest, the study involved a screening process where research staff conducted phone calls to assess eligibility. Several caregivers were excluded for reasons such as not providing sufficient care hours, lacking internet access, currently engaging in other support programs, or no diagnosis of Alzheimer's disease or related dementia.
Period: Overall Study
Arm/Group | GamePlan4Care (GP4C) | Resources4Care (R4C)
Started | 120 | 120
Completed | 79 | 88
Not Completed | 41 | 32
Not completed — Lost to Follow-up | 25 | 23
Not completed — Withdrawal by Subject | 15 | 9
Not completed — Discontinued | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GamePlan4Care (GP4C) | Resources4Care (R4C) | Total
Number analyzed (Participants) | 120 | 120 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.79 (12.83) | 64.73 (11.28) | 64.76 (12.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 95 | 193
  Male | 22 | 25 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 21 | 32
  Not Hispanic or Latino | 109 | 99 | 208
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 8 | 17
  White | 101 | 101 | 202
  More than one race | 10 | 11 | 21
  Unknown or Not Reported | 0 | 0 | 0
AD8 - Ascertain Dementia 8 [Mean (Standard Deviation); unit: Score on a Scale] — AD8 is an 8-question interview using a yes/no scoring system. The informant (i.e, family caregiver) is asked if there have been changes in areas of cognition and functioning including memory, orientation, executive function and interest in activities. The final score is a sum of the number items marked "Yes, A change" for a total potential score of 8. A score from 0 or 1 equals normal cognition. A score of 2 or greater demonstrates cognitive impairment is likely present.
  Score on a Scale | 7.44 (0.97) | 7.63 (0.74) | 7.54 (0.97)
Neuropsychiatric Inventory-Questionnaire (NPI-Q) Behavior [Mean (Standard Deviation); unit: Score on Scale] — The NPI-Q measures the presence, severity and distress ratings of 12 neuropsychiatric symptoms in patients with dementia. Each item asks the presence (1=yes, 0=no), severity (1=mild, 2=moderate, 3=severe), and caregiving distress (0=not at all; 5=extreme or very severe). NPI-Q behaviors was scored by the total sum of symptoms present (0=none at all and 12=all symptoms present).
  Score on Scale | 6.98 (2.74) | 7.04 (2.63) | 7.01 (2.68)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Caregiving Burden at 6 Months
Description: A 12-item version of the Zarit Caregiver Burden Interview. The Zarit Caregiver Burden Interview (ZBI) is an assessment tool for evaluating caregiver burden. The ZBI consists of 12 items representing a statement related to some aspect of perceived burden. Respondents (i.e., caregivers) rate each item ranging 0 (=never) to 4 (=nearly always). Total ZBI score is the summation of 12 items ranging from 0 to 48. Higher scores indicate greater burden.
Time Frame: Baseline and six months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GamePlan4Care (GP4C) | Resources4Care (R4C)
Number analyzed (Participants) | 79 | 88
score on a scale | -3.00 (6.01) | -2.75 (5.82)

2. Primary Outcome: Change From Baseline Depression at 6 Months
Description: Levels of depressed symptoms:
  A 10-item Center for Epidemiological Studies Depression Scale (CES-D) is scored from zero (= rarely or none of the time) to three (= most or all of the time). Two items are reverse scored. The total score ranges from zero to 30 indicating that higher scores are higher levels of depressive symptoms.
Time Frame: Baseline and six months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GamePlan4Care (GP4C) | Resources4Care (R4C)
Number analyzed (Participants) | 79 | 88
score on a scale | -1.57 (5.97) | -0.57 (5.43)

3. Primary Outcome: Change From Baseline Social Support at 6 Months
Description: Assessment of availability of support and satisfaction with support from others:
  Two subscales of the Social Provisions Scale (SPS), Reliable Alliance and Guidance, assessed the availability of social support and satisfaction with support received from others. Each subscale has four items. Each question is scored from one (=strongly disagree) to four (=strongly agree). Each subscale contains two questions that are reverse-scored. Ranging from four to 16, the higher total scores indicate higher levels of reliable alliance and guidance.
Time Frame: Baseline and six months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GamePlan4Care (GP4C) | Resources4Care (R4C)
Number analyzed (Participants) | 79 | 88
score on a scale
  SPS Reliable Alliance | 0.13 (2.56) | 0.01 (2.51)
  SPS Guidance | 0.42 (1.96) | 0.46 (2.33)

4. Secondary Outcome: Change From Baseline Caregiver Stress at 6 Months
Description: Assessment of levels of stress:
  Perceived Stress Scale (PSS) was used to assess the degree of stress individuals experienced, using 10 items. Each item is scored from zero to four, with a total score range of zero to 40. Four items were scored reversely. Higher total scores indicate greater perceived stress.
Time Frame: Baseline and six months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GamePlan4Care (GP4C) | Resources4Care (R4C)
Number analyzed (Participants) | 79 | 88
score on a scale | -1.41 (6.33) | -1.22 (5.64)

5. Secondary Outcome: Change From Baseline Reported Positive Aspects of Caregiving at 6 Months
Description: Assessment of favorable aspects of caregiving experiences:
  The PAC was measured with 11 items of the favorable aspects of caregiving experience. Each question is scored from zero to four with a total score ranging from zero to 44. Higher scores indicate higher levels of positive feelings from caregiving.
Time Frame: Baseline and six months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GamePlan4Care (GP4C) | Resources4Care (R4C)
Number analyzed (Participants) | 79 | 88
score on a scale | 1.95 (7.42) | 1.35 (5.75)

6. Secondary Outcome: Change From Baseline Neuropsychiatric Symptoms in Care-recipient/Corresponding Caregiver Distress at 6 Months
Description: Presence and severity of neuropsychiatric symptoms and levels of relevant caregiving distress :
  The NPI-Q measures the presence, severity and distress ratings of 12 neuropsychiatric symptoms in patients with dementia. Presence of each symptom and distress ratings for each symptom are reported as well as the total sum of dementia behaviors and distress scores for each symptom. Each dementia behavior was scored as a binary change score (yes/no). Distress is scored from zero to five with higher scores indicating higher levels of distress.
Time Frame: At Baseline and 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GamePlan4Care (GP4C) | Resources4Care (R4C)
Number analyzed (Participants) | 79 | 88
score on a scale | -2.62 (8.83) | -1.53 (7.50)

ADVERSE EVENTS:
Time Frame: Adverse event data for the participant was collected through study completion, an average of 1 year. This timeframe encompassed the duration from the start of participant enrollment through the six-month follow-up assessments, allowing for the monitoring of any adverse events related to the interventions.
Arm/Group | GamePlan4Care (GP4C) | Resources4Care (R4C)
All-Cause Mortality (participants affected / at risk) | 0/120 | 0/120
Serious Adverse Events (participants affected / at risk) | 0/120 | 0/120
Other Adverse Events (participants affected / at risk) | 0/120 | 0/120

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-01-11): https://cdn.clinicaltrials.gov/large-docs/98/NCT04540198/Prot_001.pdf
  • Statistical Analysis Plan (2025-04-21): https://cdn.clinicaltrials.gov/large-docs/98/NCT04540198/SAP_002.pdf